CLINICAL TRIAL: NCT01225913
Title: Evaluation of Mechanism(s)Limiting Expiratory Airflow in Chronic, Stable Asthmatics Who Are Non-smokers
Brief Title: Mechanism(s) of Airflow Limitation During Exacerbation of Asthma
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Gelb, Arthur F., M.D. (Individual)
Responsible Party: Principal Investigator, Arthur F Gelb MD, Principal Investigator, Gelb, Arthur F., M.D.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20070934A; NCT01225900 (obsolete NCT alias)
Record Dates: First submitted 2010-10-19; First posted 2010-10-21 (Estimated); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Asthma
Keywords: asthma; lung function; inflammation
MeSH Terms: conditions — Asthma; Inflammation | interventions — Fluticasone; Salmeterol Xinafoate; Budesonide; Formoterol Fumarate; Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Intervention Model Description: To Better Understand the Mechanism(s) of Airflow Limitation During Exacerbation of Asthma
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Asthma observational study arm (Other): Asthmatics in this arm may be on varying dose of inhaled fluticasone 100-500mcg/salmeterol 50mcg bid via Advair MDI or equivalent dose via Diskus bid or Symbicort (budesonide 80-160mcg/formoterol 4.5mcg bid)or Dulera 100-200mcg mometasone/5 mcg formoterol bid, tiotropium 18mcg capsule daily. This is an observational study and additional pharmacologic intervention may include antibiotic and tapering doses of corticosteroids.
  Interventions: Drug: fluticasone/salmeterol in all asthmatics; Drug: budesonide/formoterol or fluticasone/salmeterol in all asthmatics

INTERVENTIONS:
Drug: fluticasone/salmeterol in all asthmatics — budesonide 80ug/formoterol 4.5ug, 2 inhalations bid X 20-60 days or fluticasone 100ug/salmeterol 50ug, 1 inhalation bid X 20-60 days
  Other Names: symbicort 80/4.5; advair 100/50 or 250/50 or 500/50 bid
Drug: budesonide/formoterol or fluticasone/salmeterol in all asthmatics — budesonide 160ug/formoterol 4.5ug, 2 inhalations bid or fluticasone 250ug/salmeterol 50ug, 1 inhalations bid
  Other Names: symbicort 160/4.5; advair 250/50

SUMMARY:
The purpose of this study is to evaluate the site and mechanisms responsible for expiratory airflow limitation in chronic, treated, non-smoking, stable asthmatics with moderate to severe persistent expiratory airflow obstruction. Treatment will include inhaled corticosteroids and long acting beta2agonists. The investigators are interested in determining whether the large and/or small airways are the predominant site of airflow limitation. The investigators are also interested in determining whether intrinsic small airways obstruction and/or loss of lung elastic recoil is responsible for expiratory airflow limitation. The investigators are also interested to evaluate the role of varying doses of inhaled corticosteroids to suppress large and small airway inflammation using exhaled nitric oxide as surrogate markers of inflammation. For comparison purposes, spirometry and measurements of exhaled nitric oxide will also be obtained if possible during a naturally occurring exacerbation of asthma.

DETAILED DESCRIPTION:
In addition we will also obtain above studies in asthmatics during naturally occuring exacerbation of asthma and following treatment. If available, results of lung function studies including measurements of lung elastic recoil will be compared to pathologic analyses of formalin fixed, air inflated lungs obtained at autopsy in asthmatics who die from asthma related or non-asthma related death. This kind of lung structure-function study will provide potential mechanism(s) to explain the loss of lung elastic recoil in acute and chronic asthmatics who are non-smokers. We will also obtain voxel quantification of high resolution thin section CT of lung obtained without IV contrast. Also, we will use fiberoptic bronchoscopy to obtain optical coherence tomography in stable asthmatics with mild to moderate to severe expiratory airflow limitation to assess integrity of the lung parenchyma.

ELIGIBILITY:
Inclusion Criteria:

* Current non-smoking (<10 pack yr smoking history)
* Stable, treated asthmatics
* Age 10-80 yr
* post 180ug albuterol by MDI: FEV 1/FVC < 70% and FEV 1 <80% predicted

Exclusion Criteria:

* Pregnancy

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-10; Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Exhaled nitric oxide | 20-60 days
  evaluate the role of inhaled corticosteroid on exhaled nitric oxide production in large airways and peripheral small airways/alveoli

SECONDARY OUTCOMES:
Mechanism(s) of expiratory airflow limitation | 1 to 5 years
  loss of lung elastic recoil vs intrinsic airway obstruction
Presence of unsuspected emphysema by autopsy or explanted lung | 1-5 years
  Analysis of lungs obtained at autopsy or explanted lung for extent of emphysema

CONTACTS AND LOCATIONS:
Overall Officials: Arthur F Gelb, MD, Principal Investigator — Arthur F Gelb Medical Corporation
Locations (1):
- Arthur F Gelb Medical Corporation, Lakewood, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gelb AF, Zamel N. Unsuspected pseudophysiologic emphysema in chronic persistent asthma. Am J Respir Crit Care Med. 2000 Nov;162(5):1778-82. doi: 10.1164/ajrccm.162.5.2001037. PMID 11069812
- [Background] Gelb AF, Licuanan J, Shinar CM, Zamel N. Unsuspected loss of lung elastic recoil in chronic persistent asthma. Chest. 2002 Mar;121(3):715-21. doi: 10.1378/chest.121.3.715. PMID 11888951
- [Background] Gelb AF, Gutierrez CA, Weisman IM, Newsom R, Taylor CF, Zamel N. Simplified detection of dynamic hyperinflation. Chest. 2004 Dec;126(6):1855-60. doi: 10.1378/chest.126.6.1855. PMID 15596684
- [Background] Gelb AF, Flynn Taylor C, Shinar CM, Gutierrez C, Zamel N. Role of spirometry and exhaled nitric oxide to predict exacerbations in treated asthmatics. Chest. 2006 Jun;129(6):1492-9. doi: 10.1378/chest.129.6.1492. PMID 16778266
- [Background] Gelb AF, Taylor CF, Nussbaum E, Gutierrez C, Schein A, Shinar CM, Schein MJ, Epstein JD, Zamel N. Alveolar and airway sites of nitric oxide inflammation in treated asthma. Am J Respir Crit Care Med. 2004 Oct 1;170(7):737-41. doi: 10.1164/rccm.200403-408OC. Epub 2004 Jun 30. PMID 15229098
- [Background] Gelb AF, Zamel N, Krishnan A. Physiologic similarities and differences between asthma and chronic obstructive pulmonary disease. Curr Opin Pulm Med. 2008 Jan;14(1):24-30. doi: 10.1097/MCP.0b013e3282f197df. PMID 18043272
- [Background] Gelb AF, Yamamoto A, Verbeken EK, Schein MJ, Moridzadeh R, Tran D, Fraser C, Barbers R, Elatre W, Koss MN, Glassy EF, Nadel JA. Further Studies of Unsuspected Emphysema in Nonsmoking Patients With Asthma With Persistent Expiratory Airflow Obstruction. Chest. 2018 Mar;153(3):618-629. doi: 10.1016/j.chest.2017.11.016. Epub 2017 Nov 29. PMID 29197547
- [Result] Gelb AF, Moridzadeh R, Singh DH, Fraser C, George SC. In moderate-to-severe asthma patients monitoring exhaled nitric oxide during exacerbation is not a good predictor of spirometric response to oral corticosteroid. J Allergy Clin Immunol. 2012 Jun;129(6):1491-8. doi: 10.1016/j.jaci.2012.03.036. Epub 2012 May 2. PMID 22560478
- [Result] Gelb AF, Yamamoto A, Mauad T, Kollin J, Schein MJ, Nadel JA. Unsuspected mild emphysema in nonsmoking patients with chronic asthma with persistent airway obstruction. J Allergy Clin Immunol. 2014 Jan;133(1):263-5.e1-3. doi: 10.1016/j.jaci.2013.09.045. Epub 2013 Nov 28. No abstract available. PMID 24290280
- [Result] Gelb AF, Singh DH, Moridzadeh R, Fraser C, Tran D, Verbanck S, George SC. Age-stratified comparison of large and peripheral airway/alveolar nitric oxide levels in children and young adults. J Allergy Clin Immunol. 2013 Nov;132(5):1222-4. doi: 10.1016/j.jaci.2013.05.045. Epub 2013 Aug 6. No abstract available. PMID 23932460
- [Result] Senhorini A, Ferreira DS, Shiang C, Silva LF, Dolhnikoff M, Gelb AF, Mauad T. Airway dimensions in fatal asthma and fatal COPD: overlap in older patients. COPD. 2013 Jun;10(3):348-56. doi: 10.3109/15412555.2012.752806. Epub 2013 Mar 28. PMID 23537051
- [Result] Gelb AF, Yamamoto A, Verbeken EK, Nadel JA. Unraveling the Pathophysiology of the Asthma-COPD Overlap Syndrome: Unsuspected Mild Centrilobular Emphysema Is Responsible for Loss of Lung Elastic Recoil in Never Smokers With Asthma With Persistent Expiratory Airflow Limitation. Chest. 2015 Aug;148(2):313-320. doi: 10.1378/chest.14-2483. PMID 25950858
- [Result] Gelb AF, Christenson SA, Nadel JA. Understanding the pathophysiology of the asthma-chronic obstructive pulmonary disease overlap syndrome. Curr Opin Pulm Med. 2016 Mar;22(2):100-5. doi: 10.1097/MCP.0000000000000236. PMID 26717511
- [Result] Gelb AF, Nadel JA. Understanding the pathophysiology of the asthma-chronic obstructive pulmonary disease overlap syndrome. J Allergy Clin Immunol. 2015 Sep;136(3):553-5. doi: 10.1016/j.jaci.2015.06.013. No abstract available. PMID 26343939